CLINICAL TRIAL: NCT00307177
Title: Evaluation of the Reactogenicity and Immunogenicity of Different Doses of Trivalent Baculovirus-expressed Influenza HA Vaccine in Adults With Non-Hodgkin's B-cell Lymphoma: A Phase II, Double-Blind Pilot Study
Brief Title: Trivalent Baculovirus-expressed Influenza HA Vaccine in Adults With Non-Hodgkin's B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-036
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2006-11

CONDITIONS: Influenza
Keywords: influenza vaccine, baculovirus, immunogenicity, lymphoma
MeSH Terms: conditions — Influenza, Human; Lymphoma | interventions — trivalent baculovirus-expressed influenza-virus hemagglutinin vaccine

ARMS (4):
- Arm D (Experimental): 25 subjects receive Recombinant rHA0 vaccine at 135 mcg per rHA0, via IM injection on Day 0
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- Arm C (Experimental): 25 subjects receive Recombinant rHA0 vaccine at 45 mcg per rHA0, via IM injection on Day 0
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- Arm B (Experimental): 25 subjects receive Recombinant rHA0 vaccine at 15 mcg per rHA0, via IM injection on Day 0
  Interventions: Biological: Trivalent Baculovirus-expressed Influenza HA vaccine
- Arm A (Active Comparator): 25 subjects receive Standard TIV at 15 mcg HA per virus, in a total volume of 0.5 mL, by deep intramuscular (IM) injection on Day 0
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Standard Trivalent inactivated influenza vaccine, licensed. Arm A receives standard dose of 15 mcg IM on day 0.
  Arms: Arm A
Biological: Trivalent Baculovirus-expressed Influenza HA vaccine — Trivalent Baculovirus-expressed influenza HA vaccine (Recombinant rHA0): Arms B, C and D receive 15 mcg, 45 mcg or 135 mcg IM dose on Day 0.
  Arms: Arm B; Arm C; Arm D

SUMMARY:
The purpose of this research is to compare reactions and antibody responses following receipt of different doses of the experimental influenza vaccine or standard influenza vaccine.

DETAILED DESCRIPTION:
Influenza is a common respiratory infection caused by viruses. Epidemics of influenza occur each winter and are responsible for more than 20,000 deaths each year in the United States. Most of these deaths occur among elderly persons and among people of all ages who suffer from a chronic disease. Standard influenza vaccines may not be as effective at protecting cancer patients as the general population from getting influenza. This research study will test an experimental influenza vaccine consisting of the important flu virus protein that stimulates protection. It is produced by genetic techniques in cultured cells and allows higher doses of the protein to be used. Influenza vaccines made this way have been given to humans in the past and the vaccine was well tolerated. It is expected that higher doses of this vaccine can be given with minimal reactions, as well as whether such a vaccine stimulates higher levels of infection-fighting proteins (or antibodies) in the blood than standard doses of the licensed influenza vaccine. This study will evaluate the reactogenicity and immunogenicity of a recombiant influenza vaccine in non-Hodgkin's B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-Hodgkin's B-cell lymphoma (NHL) including follicular, large cell and Mantle cell lymphoma will be included.
* Patients in complete clinical remission and determined to have no evidence of active disease (NED).
* Ambulatory, medically stable persons; community dwelling; able to give informed consent and available for all study visits; able to understand and comply with planned study procedures; ECOG performance status less than or equal to 2.
* Medically stable subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, or hypothyroidism, but their symptoms/signs are controlled with medical therapy.
* Patients with a non-metastatic secondary solid tumor or malignancies not currently (< 3 months) being treated will be included.
* Patients greater than or equal to 18 years of age who have given informed consent and signed the IRB approved informed consent.

Exclusion Criteria:

* Patients with Hodgkin's disease, and T-cell lymphoma.
* Patients undergoing antineoplastic therapy.
* Patients who have received chemotherapy within the past 3 months.
* Individuals who were given rituximab (ibritumomab tiuxetan) in < 6 months.
* Patients receiving systemic corticosteroids and/or high-dose inhaled steroids (>800 mcg per day of beclomethasone dipropionate or equivalent).
* Splenectomized individuals will not be included.
* Known allergy to eggs or other components of vaccine (e.g., thimerosal).
* Acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses (including but not limited to the following: acute febrile illness, known chronic liver disease; significant renal disease; oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV dyspnea; unstable or progressive neurologic disorder; insulin-dependent diabetes mellitus).
* Concomitant use of investigational vaccines and/or other medications within 4 weeks prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products prior to study completion.
* Previous exposure to parenteral immunoglobulins or other blood product within 6 months prior to enrollment into the study.
* Subject is enrolled in a conflicting clinical trial.
* Use of experimental vaccines or medications within one month of study entry.
* Any acute or chronic condition which in the opinion of the investigator would render vaccination unsafe or interfere with the evaluation of response.
* Patients with a known history or risk factors (IV drug abuse or casual sex within the past year) of Hepatitis B, Hepatitis C, or Human Immunodeficeincy Virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States